CLINICAL TRIAL: NCT03104023
Title: Influence of Staple Line Inversion vs Buttressing on Postoperative Nausea or Vomits After Laparoscopic Sleeve Gastrectomy (LSG)
Brief Title: Staple Line Inversion vs Buttressing on Postoperative Vomits After LSG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Head of Bariatric Surgery Unit. Hospital general Elche, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HGUE 2016-33
Record Dates: First submitted 2017-03-24; First posted 2017-04-07 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-03

CONDITIONS: Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staple line inversion (Active Comparator): Patients will undergo a staple line inversion with a a running suture of Polypropylene 2/0.
  Interventions: Procedure: Staple line inversion
- Staple line buttressing (Experimental): The gastric section will be performed with preloaded buttress material .
  Interventions: Combination Product: Staple line buttressing

INTERVENTIONS:
Procedure: Staple line inversion — A staple line inversion will be performed with a running suture of Polypropylene 2/0
  Arms: Staple line inversion
Combination Product: Staple line buttressing — The gastric section will be performed with a stapler with preloaded buttress material
  Arms: Staple line buttressing

SUMMARY:
Patients undergoing laparoscopic sleeve gastrectomy will be randomized into 2 groups. In one group, a staple line inversion with a running suture of Polypropylene will be performed. In the second group, the gastric section will be performed with a stapler with preloaded buttress material

Postoperative nausea and vomits during the first 24 hours will be investigated.

DETAILED DESCRIPTION:
Patients undergoing laparoscopic sleeve gastrectomy as bariatric procedure will be randomized into 2 groups. In one group after the stapling and section of the stomach with stapling devices (EndoGIA, Covidien, USA), a staple line inversion with hemostatic and aims will be performed. Staple line inversion will be performed with a running suture of Polypropylene 2/0. In the second group, the gastric section will be performed with a stapler with preloaded buttress material (EndoGIA with reinforced reload, Covidien, USA).

Postoperative nausea and vomits during the first 24 hours after surgery will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40
* BMI>35 with obesity-related comorbidities

Exclusion Criteria:

* Patients undergoing other bariatric techniques than sleeve gastrectomy
* Laparotomic approach

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomits | 24 hours after surgery
  Postoperative nausea and vomits will be measured using the postoperative nausea and vomiting intensity scale, described by Wengritzky et al (Br J Anaesth 2010;104:158-166). In this scale, the number of vomits are quantified, the frequence of nausea and if it is constant or varying are determined, and the duration of the feeling of nausea is established.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, Principal Investigator — Hospital general Elche
Locations (1):
- Hospital general Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No